CLINICAL TRIAL: NCT06367023
Title: Effectiveness of Brahma Kumaris Raja Yoga Meditation on Quality of Life of Youth Residing in the Deaddiction Center of Biratnagar
Brief Title: Effectiveness of Brahma Kumaris Raja Yoga Meditation on Quality of Life of Youth in the Deaddiction Center of Biratnagar
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Manipur International University (Other)
Collaborators: Brahmakumaris (Unknown)
Responsible Party: Principal Investigator, Rajiv Ranjan Karn, Principal Investigator, Manipur International University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 32-2024
Record Dates: First submitted 2024-03-29; First posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Prevalence; Depression; Happiness; Quality of Life; Anxiety
Keywords: Anxiety; meditation; drug addiction
MeSH Terms: conditions — Depression; Anxiety Disorders; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rajyoga Meditation Practice (Experimental): Rajyoga Meditation Intervention: 3 months, For 6 days one hour per day Rajyoga meditation basic course will be provided, followed by 1 hour daily spiritual lesson, Positive thinking and motivation classes will be provided to the intervention group where 1. Initiation - In this stage, thoughts in the mind, come in randomly, 2. Concentration - He now, converts all negative thoughts with positive thoughts of peace, happiness, love, bliss, purity, knowledge, and power 3. Realization - This final stage involves feeling the emotions of these positive thoughts and in the control group standard treatment will be given.
  Follow-up: Follow up will be done after 1 month of discharge from the rehabilitation centers.
  Interventions: Behavioral: Rajyoga Meditation Practice
- Standard of care (No Intervention): The usual therapy of the rehabilitation center will be given for 3 months. Baseline, 3 month and follow up after 1 month will be taken

INTERVENTIONS:
Behavioral: Rajyoga Meditation Practice — The intervention will be given for 3 months, For 6 days one hour per day Rajyoga meditation basic course will be provided, followed by 1 hour daily spiritual lesson, Positive thinking and motivation classes will be provided to the intervention group and in control group standard treatment will be given.
  Arms: Rajyoga Meditation Practice

SUMMARY:
Drug addiction is a public health problem, mainly youths are involved in the addiction and the major reason were due to peer pressure. Spiritual meditation is thought to foster a deeper sense of meaning, which creates new sources of positive reinforcement, increasing motivation for alternative behavior patterns, such as entering treatment or maintaining abstinence. Cluster Randomized Control Trial will be performed for 1-year period where mixed method study design will be performed. The major variables will be Anxiety and depression score, Happiness index, Quality of life, Rate of Relapse, Age, Gender, Occupation, Education, Income, Family Size, Family Income, Family support, Social status- High/Middle/Low, History of drug use self, Types of drugs, Duration of usage: Reason of drug use, how they have started, Amount of drugs, Frequency of use, Family history of drug use, Money spent on drugs per month. A modified validated Questionnaire will be used. CRCT will be done by CONSORT Guidelines. A total of 160 samples will be taken, (40 from each center, two were given Meditation intervention and 80 were given standard treatment as a control group) and 16 qualitative interviews will be taken (4 from each center). The intervention will be given for 3 months, for 6 days one hour per day Rajyoga meditation basic course will be provided, followed by a 1-hour daily spiritual lesson, Positive thinking and motivation classes will be provided to the intervention group, and in the control group standard treatment will be given. Follow-up will be done after 1 month of discharge from the rehabilitation centers. Ethical clearance will be taken from the Ethical Review Board (ERB) of the Nepal Health Research Council (NHRC). This study will be useful for developing policy and practice in rehabilitation centers to apply the technique of Rajyoga Meditation in relapse prevention.

DETAILED DESCRIPTION:
Introduction Globally 2.4 million people were current drinkers. In 2020, 22.3% of the world's population used tobacco: 36.7% of men and 7.8% of women. Around 80% of the 1.3 billion tobacco users worldwide live in low- and middle-income countries.

The problem of Substance use/drug use in Nepali society has traditionally been dominated by cannabis and opioids. But this list has now expanded to include 'hard drugs' like the South Asian cocktail which is a mixture of opioids, benzodiazepine, and antihistamines. Heroin (Diacetyl morphine), injectable buprenorphine, and pharmaceutical opioids is currently known to be frequently used opioids in Nepal.

The reason for starting drug use was mainly due to peer pressure 89%, recreation 72%, and curiosity 62%. Fifteen percent of the drug users suffer from Hepatitis B/C, 36% are from lower secondary education and 39% of drug users are unemployed. Due to this various personal, professional, and social problem arises. The drug users have expectations from the government 39% said cross-border screening and checking to reduce drug use and 47% said there should be employment opportunities to improve the lives of drug users.

Despite this huge problem only one in seven people with drug users receive treatment.

Different rehabilitation centers in Nepal are led by NGOs and some are privately run.

Rehabilitation centers help to enhance self-confidence among drug abusers and enable them to dislike drugs, to create public awareness in society via various programs showing the ill effects of the drugs. It helps to decrease the criminal activities caused by drug addiction, to decrease the consumption of the drugs by the users, and also to control the import and export of drugs.

Spiritual meditation is thought to foster a deeper sense of meaning, which creates new sources of positive reinforcement, increasing motivation for alternative behavior patterns, such as entering treatment or maintaining abstinence.

Meditation techniques may offer additive benefits to standard outpatient treatment compared to standard treatment alone, specifically in maintaining abstinence.

Short-term spiritual-based relaxation therapy (Rajyoga meditation) was highly effective in causing earlier relief in chronic tension headaches. If we can change our thinking, ahara, vihara, then we will be able to change the quality of life.

Rationale of the study: Youths are the future of the Nation. The literature shows that spirituality and Brahmakumaris Raja Yoga meditation is effective in reducing anxiety and helpful for Coronary heart diseases. There are very few studies that show the Impact of yoga and physical exercise on psychological wellbeing among substance abusers but very limited studies show the effects of Raja Yoga meditation to improve relapse prevention in Nepal. Hence the aim to measure the effects of Raja Yoga Meditation among youths who are residing in rehabilitation centers of Biratnagar. These findings will help develop a policy to implement spiritual-based practice to improve the quality of life and reduce relapse prevention.

Hypothesis H0: There is no difference in relapse prevention between Rajyoga meditation along with rehabilitation center treatment and rehabilitation center treatment alone.

4. General Objective To find out the Prevalence of anxiety, depression score, happiness index, and quality of life among people residing in rehabilitation centers To explore the life experiences of youth residing in the rehabilitation centers before and after the meditation program.

To find out the effect of Brahma Kumaris Raja Yoga meditation on relapse prevention and improving the quality of life of youth residing in the selected Rehabilitation center of Biratnagar.

Study Variables Outcome variables Primary outcome: Depression, Anxiety and Stress Secondary outcome: Rate of Relapse Independent variables Age, Gender, Occupation, Education, Income, Family Size, Family Income, Family support

Social status- High/Middle/Low, History of drug use self, Types of drugs, Duration of usage:

Reason of drug use, How you have started, Amount of drugs, Frequency of use, Family history of drug use, Money spent on drugs per month Methodology Research Methods: Mixed Data collection: Data will be collected for baseline, after 3 months, and 1 month after discharge from the rehabilitation center, Study site and its justification: Biratnagar Metropolitan City.

Specify type of study: Cluster Randomized Controlled Trial (CRCT) Sample size: Total 409, 369+40(10% nonresponse), assuming 60% prevalence of relapse as per the study(Kabisa- 2021) For intervention 160, (40 from each center, two was given Meditation intervention and 80 were given standard treatment as control group) 16 qualitative interview will be taken (4 from each center) Sampling technique: From the list of rehabilitation centers, two rehabilitation centers will be selected randomly for the intervention group and two for the control group by lottery method.

CRCT will be done by CONSORT Guidelines. Period of study: 1 year Method of randomization: Simple randomization, the clusters will be randomized to the intervention or control arm.

Intervention: 3 months, for 6 days one hour per day Rajyoga meditation basic course will be provided, followed by one-hour daily spiritual lesson, Positive thinking and motivation classes will be provided to the intervention group where Experimental population: All youths residing in the rehabilitation center and who are under treatment of different rehabilitation centers of Biratnagar Metropolitan city.

Study unit: Individual youth residing in rehabilitation centers Inclusion criteria: Those youth more than 18 years old who had used drugs and residing in the rehabilitation center of Biratnagar and giving consent will be involved in the study.

Data collection Technique: Face-to-face interview and in-depth interviews will be used for qualitative study.

Ethical consideration: Ethical clearance will be taken from the Ethical Review Board (ERB) of Nepal Health Research Council (NHRC) and Manipur International University, Data collection tools: A modified validated Questionnaire will be used WHOQOL-SRPB field-test instrument. World Health Organization had developed the tools to measure the quality of life spirituality, religiousness, and personal beliefs (SRPB) -32 items.

The data will be categorized by Cut off-point Determinants of drug abuse A pretesting will be conducted to measure the appropriateness of the questionnaire and the time taken to complete it, Piloting: A pilot study will be done in one of the rehabilitation centers at Lahan to find out the feasibility, and acceptability of certain policies and to check whether there is any flaws.

Analysis Plan Data integration: Once both quantitative and qualitative data are analyzed separately, we will compare the results from both and tie findings together.

Expected outcome of the study The expected outcome of the effects of Brahamakumari Raj Yoga Meditation on the quality of life of youth residing in the rehabilitation center of Biratnagar include the current situation of anxiety, depression, and quality of life, and how meditation helps reduce relapse.

Significance and Contribution This study will be useful for developing policy and practice in rehabilitation centers to apply the technique of Rajyoga Meditation in relapse prevention and lead their life and health.

ELIGIBILITY:
Inclusion Criteria:

* Those youth more than 18 years old
* Who had used drugs and residing in the rehabilitation center of Biratnagar and
* Gave consent will be involved in the study.

Exclusion Criteria:

* Those having other illnesses and unable to give consent

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2024-10-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Anxiety score | 6 month
  Anxiety score before and after, lower score means healthy
Depression score | 6 month
  Depression score before and after lower score means healthy
quality of life score | 6 month
  Quality of life before and after higher score means healthy

SECONDARY OUTCOMES:
Rate of Relapse | 1 year
  After 1 year rate of relapse will be assessed number of person get relapsed

CONTACTS AND LOCATIONS:
Locations (1):
- Rehabilitation center, Biratnagar, Koshi, Nepal

IPD SHARING:
Plan to Share IPD: No
As per the request data will be shared

REFERENCES:
- [Background] Berking M, von Kanel M. [Mindfulness training as a psychotherapeutic tool. Clarification of concept, clinical application and current state of empirical research]. Psychother Psychosom Med Psychol. 2007 Mar-Apr;57(3-4):170-7. doi: 10.1055/s-2006-951956. German. PMID 17427100
- [Background] Bizzarri J, Rucci P, Vallotta A, Girelli M, Scandolari A, Zerbetto E, Sbrana A, Iagher C, Dellantonio E. Dual diagnosis and quality of life in patients in treatment for opioid dependence. Subst Use Misuse. 2005;40(12):1765-76. doi: 10.1080/10826080500260800. PMID 16419555
- [Background] Chapagain K, Rai D, Koirala B, Rauniyar GP. Exploring the Prevalence and Correlates of Substance Abuse Amongst the Adolescents of Dharan, Eastern Nepal. J Nepal Health Res Counc. 2020 Sep 8;18(2):263-267. doi: 10.33314/jnhrc.v18i2.2484. PMID 32969390
- [Background] GBD 2016 Alcohol Collaborators. Alcohol use and burden for 195 countries and territories, 1990-2016: a systematic analysis for the Global Burden of Disease Study 2016. Lancet. 2018 Sep 22;392(10152):1015-1035. doi: 10.1016/S0140-6736(18)31310-2. Epub 2018 Aug 23. PMID 30146330
- [Background] Hayes, S. C. (2015). The Act in Context: The Canonical Papers of Steven C. Hayes. Routledge.